CLINICAL TRIAL: NCT02985840
Title: Ondansetron Versus Dexamethasone/Ondansetron to Treat Acute Nausea in the Emergency Department
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Unable to access EMR for patients enrolled prior to 8/2015 for data collection
Sponsor: OhioHealth (Other)
Responsible Party: Principal Investigator, Andrew Little, Attending Physician, OhioHealth
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1066755 (13-0056)
Record Dates: First submitted 2016-10-30; First posted 2016-12-07 (Estimated); Results first posted 2018-09-26 (Actual); Last update posted 2018-09-26 (Actual); Status verified 2018-08

CONDITIONS: Nausea; Abdominal Pain
Keywords: ondansetron; dexamethasone
MeSH Terms: conditions — Nausea; Abdominal Pain | interventions — Ondansetron; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ondansetron (Active Comparator): Ondansetron (4 mg) followed by two 5 ml normal saline flush
  Interventions: Drug: Ondansetron
- Ondansetron plus dexamethasone (Experimental): Ondansetron (4 mg), followed by dexamethasone (4 mg), followed by a single 5 ml normal saline flush
  Interventions: Drug: Ondansetron; Drug: Dexamethasone

INTERVENTIONS:
Drug: Ondansetron — Patients receive intravenous ondansetron (4mg) followed by two 5ml normal saline flushes
  Other Names: Zofran
Drug: Dexamethasone — Patients receive intravenous ondansetron(4mg) followed by intravenous dexamethasone (4mg), followed by a single 5ml normal saline flush
  Other Names: Decadron
  Arms: Ondansetron plus dexamethasone

SUMMARY:
Nausea is a common complaint in patients who present to the emergency department (ED). Although the number of conditions that can present with nausea are numerous, the mainstay of treatment has become intravenous ondansetron (Zofran), not only due to its rapid onset but also its availability. One of the major drawbacks to using this form is that it often needs to be redosed. This study aims to compare intravenous (IV) ondansetron alone versus IV ondansetron given with IV dexamethasone (Decadron) as another viable option when treating patients with nausea in the emergency department.

Previous studies in patients undergoing surgical procedures have shown that when IV dexamethasone is given with IV ondansetron to post-operative patients they have less nausea and vomiting than ondansetron alone, and were even found to show decreased post-operative pain associated with nausea. It has also been shown to decrease the need to re-dose antiemetic medication. Although this combination has not been tested in the emergency department it is believed by these investigators that the additional use of dexamethasone may decrease the need to use repeated doses of ondansetron.

The investigators believe this may change the way physicians currently approach the nauseated patient in regards to treatment. That rather than possibly giving multiple doses of one medication over and over to reduce a patient's nausea, physicians can give two medications together at one time. The investigators hope to demonstrate that by giving intravenous dexamethasone and ondansetron together, it may be possible to reduce the number of patients who need additional doses of nausea medication.

DETAILED DESCRIPTION:
Nausea is a common complaint in patients who present to the emergency department (ED). Although the number of conditions that can present with nausea are numerous, the mainstay of treatment has become intravenous ondansetron (Zofran), not only due to its rapid onset but also its availability. One of the major drawbacks to using this form is that it often needs to be redosed. This study aims to compare intravenous (IV) ondansetron alone versus IV ondansetron given with IV dexamethasone (Decadron) as another viable option when treating patients with nausea in the emergency department.

ELIGIBILITY:
Inclusion Criteria:

* Chief Complaint of nausea or abdominal pain with nausea
* Inability to tolerate oral nausea medication
* Patients with a negative pregnancy test

Exclusion Criteria:

* Patients younger than 18 years of age
* Patient's chief complaint includes headache, chest pain, or dizziness
* Patients with whom there are contraindications to using the studied medicine (allergies, known adrenal disease)
* Blood sugar greater than 300
* Non-English speaking subjects

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2014-01-28 (Actual); Primary Completion 2016-11-15 (Actual); Study Completion 2016-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Little, D.O., Principal Investigator — Attending Physician
Locations (1):
- OhioHealth Doctors Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ondansetron | Ondansetron Plus Dexamethasone
Started | 64 | 63
Completed | 64 | 63
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ondansetron | Ondansetron Plus Dexamethasone | Total
Number analyzed (Participants) | 64 | 63 | 127
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.77 (11.46) | 34.65 (12.75) | 35.21 (12.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 43 | 88
  Male | 19 | 20 | 39
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 64 | 63 | 127

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Need for Additional Nausea Medications
Description: Effectiveness of intervention will be assessed by the need for additional medications via chart review
Time Frame: 1 hour post intervention
Population: Evaluation of this outcome (need for additional medications within 1 hr of intervention) required additional chart review, which was not performed. As such, this outcome was not collected or analyzed, and cannot be reported.
Arm/Group | Ondansetron | Ondansetron Plus Dexamethasone
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Number of Participants With Resolution of Nausea and Abdominal Pain Symptoms
Description: Effectiveness of intervention will be assessed by the resolution of symptoms via chart review
Time Frame: 1 hour post intervention
Population: Evaluation of this outcome (resolution of symptoms following intervention) required additional chart review, which was not collected. As such, this outcome was not collected or analyzed, and cannot be reported.
Arm/Group | Ondansetron | Ondansetron Plus Dexamethasone
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Participants are in the study from time of enrollment until they are discharged from the emergency department. Adverse Events are collected during study enrollment. Incidence of adverse events were collected throughout the patient admission to the Emergency Department, per standard care procedures.
Description: Adverse event reporting followed local, state and federal regulations.
Arm/Group | Ondansetron | Ondansetron Plus Dexamethasone
All-Cause Mortality (participants affected / at risk) | 0/64 | 0/63
Serious Adverse Events (participants affected / at risk) | 0/64 | 0/63
Other Adverse Events (participants affected / at risk) | 0/64 | 0/63

LIMITATIONS AND CAVEATS:
Due to the transfer of electronic medical record systems, investigators were unable to access data from patients who were enrolled prior to August 2015 for the retrospective chart review component of this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes